CLINICAL TRIAL: NCT04770883
Title: Phenotyping and Treatment of Primary Health Care IBS Patients. A Randomized Controlled Trial
Brief Title: Psychological and Dietary Treatment in IBS
Acronym: ROLIBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 261771
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Cognitive Behavioral Therapy; Diet Therapy; Low FODMAP Diet; Internet Based Cognitive Behavioral Therapy; Psychological Therapy; Psychological Parameters; Phenotyping of Irritable Bowel Syndrome Patients; Gastrointestinal Symptoms; Quality of Life; Irritable Bowel Syndrome Symptom Severity
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: The study design is an open labelled, randomized, controlled clinical trial, with a ratio 2:2:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet based cognitive behavioral therapy group (Experimental): 80 patients will be randomized to receive iCBT. Psychological therapy is effective in IBS patients. The treatment takes 10 weeks and is divided into five successive steps. Patients have to report that they have worked through a treatment step to get access to the next. The patients will be encouraged to work through steps 1-4 during the first half of the treatment and to spend the latter half of the treatment on step 5, in which exposure exercises are introduced. A psychologist/CBT therapist will manage the online therapeutic contact with the patients.
  Interventions: Behavioral: Internet based cognitive behavioral therapy.
- Low FODMAP group (Experimental): 80 patients will then be randomized to receive Low FODMAP diet. FODMAPs (Fermentable Oligosaccharides, Disaccharides, Monosaccharides And Polyols) are poorly absorbed short-chain carbohydrates including fructose (in excess of glucose), lactose, polyols, fructans and galacto-oligosaccharides. The concept of considering all these molecules collectively as a treatment for IBS is relatively new. Understanding of FODMAPs comprises mechanisms of action such as luminal distension from their osmotic effect and rapid fermentation to hydrogen. These findings have led to increased application of the low FODMAP diet to manage IBS symptoms. Treatment will undergo 10 weeks supervised monotherapy with low FODMAP diet. This will be done with the help of professional dieticians in Örebro region, who will meet the patients and inform them how this diet works as well as follow up.
  Interventions: Dietary Supplement: Low FODMAP diet therapy
- Control group (Active Comparator): The control Group (40 patients) will wait for 10 weeks before being randomised to treatment with either iCBT or low FODMAP diet.
  Interventions: Behavioral: Internet based cognitive behavioral therapy.; Dietary Supplement: Low FODMAP diet therapy

INTERVENTIONS:
Behavioral: Internet based cognitive behavioral therapy. — Patients will receive iCBT for 10 weeks, divided into five successive steps. The iCBT will be guided by online therapists and emphasizes acceptance of symptoms through exposure training. Patients have to report that they have worked through a treatment step to get access to the next. Patients will be encouraged to work through steps 1-4 during the first half of the treatment and to spend the latter half on step 5, in which exposure exercises will be introduced. The treatment aims to break the vicious cycle between avoidance behavior, symptom severity and functional impairment.
  Arms: Control group; Internet based cognitive behavioral therapy group
Dietary Supplement: Low FODMAP diet therapy — Patients will receive 10 weeks of standardized treatment with low FODMAP diet consisting of 3 stages: FODMAP restriction; FODMAP reintroduction and FODMAP personalization. These stages will be covered in at least three appointments by primary care dieticians in Region Örebro County.
  Arms: Control group; Low FODMAP group

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common functional gastrointestinal (GI) condition which is strongly associated with dietary and psychosocial factors. Management of IBS remains challenging for primary health care.

The aim is to perform a comprehensive phenotyping of patients with IBS within the primary health care in Region Örebro County, Sweden. Following this phenotyping, the investigators will perform a prospective randomized controlled trial of two different treatments versus control as described below. Subsequently, the investigators want to evaluate the result of the treatments in order to see whether the presence of a certain phenotype can predict the efficacy of different treatments.

Our hypothesis is that the presence of certain baseline symptom characteristics in patients with IBS can predict how effective internet based cognitive behavioral therapy (iCBT) and low FODMAP (low Fermentable Oligosaccharides, Disaccharides, Monosaccharides, and Polyols) treatment will be for each patient.

200 patients with IBS aged 18-65 years will be recruited from the primary health care in Region Örebro County.

The study plan is structured as follows:

1. Phenotyping of IBS patients. Investigation of the correlation between different psychological parameters, IBS symptom severity and Quality of Life.
2. The effect and outcome of 10-weeks internet-based cognitive behavioral therapy (iCBT) versus control in IBS patients.
3. The effect and outcome of 10-weeks low FODMAP diet versus control in IBS patients.
4. Comparison of iCBT and low FODMAP treatment in IBS patients and identification of baseline phenotypic characteristics predicting treatment outcome for both treatments.

Stool and blood samples will be taken before and after treatment for analysis of gut microbiota, proteomics and epigenetics and to correlate these with the clinical phenotype.

All participants will undergo phenotyping regarding GI symptoms and psychological variables using questionnaires. Participants will afterwards be randomised to either 10 weeks treatment with iCBT (80 participants), low FODMAP (80 participants) or control group (40 participants) (2:2:1 randomization). The control group will wait 10 weeks before being randomised to either iCBT (20 participants) or low FODMAP (20 participants).

Significance

This study will provide effective and individualized treatment for IBS patients. This may lead to the development of a guideline to improve the effectiveness of treatment and care for patients with IBS.

DETAILED DESCRIPTION:
Part 1

Study design:

Cross-sectional observational study.

Study population:

200 IBS patients, M/F, age 18-65 years, will be recruited under a period of 4 years from the primary health care in Region Örebro County. Patients will also be recruited from the general public using websites, social media and advertisements.

Data collection:

After informed consent is signed, a doctor's assessment is made including medical history, physical examination and laboratory tests.

For assessment of the IBS symptoms but also comorbid conditions such as upper GI symptoms, somatization and psychiatric symptoms, 12 different validated questionnaires will be used to identify sub-populations (phenotypes).

All patients will be asked to fill in these questionnaires before starting, during and after treatment.

Stool and blood samples will be taken at baseline and after treatment and will be stored at a biobank for later analysis of microbiomics, proteomics and epigenetics.

Analysis:

Descriptive statistics to identify different IBS features, and Pearson's correlations to study between-person correlations in a correlation network to see which parameters correlate most with the IBS symptom scale (GSRS-IBS) and Quality of life (IBS-QoL). They will be used as the dependent variables in multiple linear regression analysis with the other parameters as independent variables.

Part 2 and 3

Study design:

Randomized controlled clinical trial.

Study population:

Patients will then be randomized to either iCBT (80 patients), Low FODMAP diet (80 patients) or control group (40 patients) (2:2:1 randomization). The control group will wait 10 weeks before being randomised to treatment with either iCBT (20 patients) or low FODMAP diet (20 patients).

Treatments:

iCBT and Low FODMAP diet (see below).

Analysis:

Treatment efficacy analysis using linear mixed models on the primary outcome measures with time as within-subject factor (random intercept random slope models) and group as between-subject factor, with the time-by-group interaction effect testing the hypothesis of a stronger response to treatment compared to waiting list control. Continuous variables will be used to maximize power. Within-person correlations between IBS features. Linear mixed models and latent class growth analysis to establish which baseline parameters of IBS predict the treatment effect on the GSRS-IBS and IBS-QoL. Cross-lagged panel models to investigate the temporal order of change in the different outcome variables, while controlling for stabilities over time and cross-sectional correlations.

Part 4

Comparison of psychological and dietary treatment in IBS patients. At this point the investigators will have 100 patients who were treated with ICBT and 100 patients who were treated with low-FODMAP diet. Treatment efficacy will be analyzed using linear mixed models on the primary outcome measures with time as within-subject factor (random intercept random slope models) and group as between-subject factor, with the time-by-group interaction effect testing the hypothesis of a stronger response to iCBT compared to low-FODMAP.

Power calculation:

It is estimated that 100 participants per group need to be included in the treatment studies and the analysis of predictors of treatment responses with regard to a dropout rate of 10% (part 2-4). For part 1, the analysis can be performed on the entire study population of 200 participants, which gives 90% power to be able to detect an effect size (Cohen's f² = 0.10) in multiple regression analysis with 9 independent variables (derived from questionnaire PHQ-9, GAD-7, PHQ-12, VSI, IBS-BRQ and NEO-FFI) predicting the severity of IBS symptoms (IBS-SSS and GSRS-IBS) and quality of life (IBS-QoL).

ELIGIBILITY:
Inclusion Criteria:

1. IBS symptom severity score of at least 175 (moderate to severe symptoms).
2. Age 18 to 65 years.

Exclusion Criteria:

1. Abnormal results on standard screening laboratory tests; this means that patients with abnormal thyroid-stimulating hormone (TSH), increased f-calprotectin or positive celiac disease serology will not be included.
2. Severe psychiatric, systemic inflammatory diseases, inflammatory bowel disease and other severe diseases such as cancer.
3. Current drug or alcohol abuse.
4. Inability to complete questionnaires in Swedish.
5. Current pharmacological treatment for their IBS symptoms, except for "over the counter" products such as loperamide or fiber.
6. Ongoing use of low FODMAP (Fermentable Mono-, di-, oligosaccharides, and polyols) diet. A current lactose free or gluten free diet will not be accepted. Earlier lactose or gluten free diet will be accepted after a wash-out period of at least 2 weeks.
7. Current psychological treatment.
8. Current psychological treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale-IBS (GSRS-IBS) | 10 weeks
  Measures disease-specific symptoms in IBS patients
The IBS quality of life questionnaire (IBS-QoL) | 10 weeks
  Assessment of disease-specific quality of Life

SECONDARY OUTCOMES:
Patient Health Questionnaire Anxiety module (GAD-7) | 10 weeks
  Measures anxiety
Patient Health Questionnaire Depression Module (PHQ-9) | 10 weeks
  Measures depressive symptoms
Patient Health Questionnaire Somatic symptom severity ('somatization') module (PHQ-12) | 10 weeks
  Measures somatic symptom severity
Visceral Sensitivity Index (VSI) questionnaire | 10 weeks
  Measures GI symptom-specific anxiety
The Irritable Bowel Syndrome-Behavioural Responses Questionnaire (IBSBRQ) | 10 weeks
  Measures treatment outcome of iCBT.
Nepean Dyspepsia Index (NDI) | 10 weeks
  Measures quality of life in functional dyspepsia
IBS severity scoring system (IBS-SSS) | 10 weeks
  Measures GI symptoms and effect of IBS on life in general
Rome IV diagnostic questionnaire | 10 weeks
  Diagnostic IBS criteria
The Neuroticism-Extraversion-Openness Five Factor Inventory-3 (NEO-FFI-3) questionnaire | 10 weeks
  Assessment of personality type based on the five-factor model: Openness, conscientiousness, extraversion, agreeableness, and neuroticism.
Bristol Stool Form Scale | 10 weeks
  Describes the stool consistency

CONTACTS AND LOCATIONS:
Locations (1):
- Skebäck primary health care center, Örebro, Sweden